CLINICAL TRIAL: NCT07066462
Title: Effect of Exercise on Human Fatigue and Performance in Healthy Individuals
Brief Title: Exercise Fatigue Prediction in Healthy Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University (Other)
Responsible Party: Principal Investigator, National Taipei University, Muhammad Adeel, DPT, Ph.D., National Taipei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ECKIRB1121004
Record Dates: First submitted 2025-06-17; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Healthy Young Adults
Keywords: Physical Fatigue Detection; Surface Electromyography (sEMG); Fatigue Monitoring; Wearable Sensors; Biosignal Analysis; Electroenchephalography (EEG); Heart rate (HR)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Protocol (Experimental): Participants in this arm will perform two physical exercises on different days while wearing sensors that measure muscle activity (sEMG), brain activity (EEG), and heart rate (HR).
  Interventions: Other: Fatigue Exercise Protocol with Biosignal Monitoring

INTERVENTIONS:
Other: Fatigue Exercise Protocol with Biosignal Monitoring — Participants will complete two fatiguing exercises, including static bicycling and dumbbell squats. During each exercise, surface electromyography (sEMG), electroencephalography (EEG), and heart rate (HR) will be recorded to analyze fatigue levels.

SUMMARY:
The goal of this research study is to develop an AI-based model to detect physical fatigue in healthy young adults. The main questions it aims to answer are:

1. Can muscle, heart, and brain signals be used to predict physical fatigue in real time?
2. How accurately can an AI model detect fatigue based on these signals?

Participants will:

* Perform moderate to high intensity physical exercises, including static bicycling and dumbbell squats, while wearing non-invasive sensors that measure muscle activity (sEMG), heart rate (HR), and brain activity (EEG).
* Before starting the exercises, participants will complete a brief warm-up session that includes stretching and mobility movements.
* Each participant undergoes two training sessions, with pre- and post-evaluations of their physical fitness status and static muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 30 years old
* Healthy college students who regularly exercise
* Participants who meet the World Health Organization (WHO) guidelines for physical activity: at least 150-300 minutes of aerobic activity per week or muscle-strengthening exercises for major muscle groups on 2 or more days per week
* Participants who provide written informed consent

Exclusion Criteria:

* Individuals younger than 18 or older than 30
* History of any metabolic, systemic, or musculoskeletal disorder
* Recent injury or surgery
* Failure to pass the pre-exercise fitness screening questionnaire (PAR-Q)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
EEG (Electroencephalography) Alpha, Beta, Delta, and Theta Band Frequency (Hz) | Two sessions: Day 1 (Cycling session) and Day 2 (Squat session)
  Relative power in the alpha (8 to 12 Hz), beta (12 to 30 Hz), delta (2 to 4 Hz), and theta (4 to 8 Hz) bands extracted from EEG signals recorded during exercise. Alpha power is associated with the onset of physical fatigue and is computed using MATLAB.
sEMG (Surface Electromyography) amplitude (μV) and median frequency (MDF) (Hz) | Two sessions: Day 1 (Cycling session) and Day 2 (Squat session)
  sEMG (microvolts) recorded from both sides of the quadriceps, hamstrings, tibialis anterior, and gastrocnemius muscles. Signal processing will be performed to compute amplitude and median frequency, assessing neuromuscular activation and fatigue during exercise.
Heart rate (HR) and Heart rate variability (HRV) | Day 1 (Cycling session) and Day 2 (Squatting session)
  Heart rate (HR) and heart rate variability (HRV) are recorded in beats per minute (bpm) throughout cycling and squat sessions. Average and peak heart rates, as well as average heart rate variability (HRV), are used to evaluate physical fatigue and cardiovascular stress.

SECONDARY OUTCOMES:
Body mass index (BMI) | Two times: before and after exercise sessions
  BMI is recorded by measuring body weight and height
Static muscle strength (N) | Two times: before and after exercise sessions
  Static muscle strength in Newton of both sides of the quadriceps, hamstrings, tibialis anterior, and gastrocnemius is recorded using a dynamometer
Borg rate of perceived exertion score (RPE) | Two sessions: Day 1 (Cycling session) and Day 2 (Squat session)
  RPE scale records physical fatigue level for two exercise sessions

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Adeel, PhD, Principal Investigator — National Taipei University
Locations (1):
- National Taipei University, Master Program in Smart Healthcare Management, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YL, Chen CC, Hsia PY, Lin SK. Relationships of Borg's RPE 6-20 scale and heart rate in dynamic and static exercises among a sample of young Taiwanese men. Percept Mot Skills. 2013 Dec;117(3):971-82. doi: 10.2466/03.08.PMS.117x32z6. PMID 24665812
- [Background] Buzsaki, G. (2006). Rhythms of the Brain: Oxford university press
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Borghini G, Vecchiato G, Toppi J, Astolfi L, Maglione A, Isabella R, Caltagirone C, Kong W, Wei D, Zhou Z, Polidori L, Vitiello S, Babiloni F. Assessment of mental fatigue during car driving by using high resolution EEG activity and neurophysiologic indices. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:6442-5. doi: 10.1109/EMBC.2012.6347469. PMID 23367404
- [Background] Bedo BLS, Pereira DR, Moraes R, Kalva-Filho CA, Will-de-Lemos T, Santiago PRP. The rapid recovery of vertical force propulsion production and postural sway after a specific fatigue protocol in female handball athletes. Gait Posture. 2020 Mar;77:52-58. doi: 10.1016/j.gaitpost.2020.01.017. Epub 2020 Jan 21. PMID 31986376
- [Background] Adeel M, Chen HC, Lin BS, Lai CH, Wu CW, Kang JH, Liou JC, Peng CW. Oxygen Consumption (VO2) and Surface Electromyography (sEMG) during Moderate-Strength Training Exercises. Int J Environ Res Public Health. 2022 Feb 16;19(4):2233. doi: 10.3390/ijerph19042233. PMID 35206420